CLINICAL TRIAL: NCT06102694
Title: Screening and Identification of Plasma Biomarkers for Early Diagnosis of Transplant-associated Thrombotic Microangiopathy Based on Proteomics and Metabolomics Techniques
Brief Title: Identification of Plasma Biomarkers for Early Diagnosis of Transplant-associated Thrombotic Microangiopathy
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QTJC2023036
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-12

CONDITIONS: Thrombotic Microangiopathies; Hematopoietic Stem Cell Transplantation
Keywords: TA-TMA; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Thrombotic Microangiopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood will be collected to reserve plasma and mononuclear cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this clinical trial is to learn about plasma biomarkers of diagnosed transplant-associated thrombotic microangiopathy (TA-TMA) in patients undergoing transplantation. The main questions it aims to answer are: whether there are molecules that can accurately diagnose and predict TA-TMA; whether the current biomarkers related to TA-TMA can well predict the occurrence and survival of TA-TMA in adult patients with malignant hematopoietic diseases, for example, acute leukemia. Participants will receive laboratory tests of peripheral blood and urine specimens related to TA-TMA at regular times after transplantation.

DETAILED DESCRIPTION:
Transplant-associated thrombotic microangiopathy (TA-TMA) is a commonly serious complication after allogeneic hematopoietic stem cell transplantation (allo-HSCT). As the diagnostic criteria are not standardized, the incidence of TA-TMA has been reported in the literature to be 0.5%-64%. TA-TMA has an insidious onset, diverse clinical manifestations, rapid progression, limited therapeutic options, and a poor prognosis, with a mortality rate of 60%-90%. The exact pathogenesis of TA-TMA is not yet fully understood. Markers of endothelial damage such as thrombomodulin (TM), plasminogen activator inhibitor-1(PAI-1), intercellular adhesion molecule-1(ICAM-1), and soluble membrane attack complex (sC5b-9) may have predictive roles, but there is a lack of large-scale prospective clinical studies to confirm it. The emergence of multi-omics technologies has brought biomarker research into the high-throughput stage. However, proteomics and metabolomics biomarkers have not been reported in TA-TMA research. In this study, the investigors will establish the first prospective study cohort for screening early warning biomarkers of TA-TMA in China, collect transplantation-related clinical data, and collect plasma serial samples from post-transplantation patients, which are expected to obtain new biomarkers that can be used in the early diagnosis of TA-TMA through the combined analysis of proteomics and metabolomics.

The contents of this study are as follows:

1. Establish the first prospective study cohort for screening TA-TMA early warning biomarkers in China. Patients will be enrolled continuously who undergo allo-HSCT in order to build a prospective study cohort to search for clinical phenotypes related to the occurrence, evolution, or prognosis of TA-TMA, and to excavate the risk factors of TA-TMA, prognostic factors, etc. Collect complete transplantation-related clinical data, and plasma serial samples at fixed testing time points. SC5b-9, urine protein to creatinine ratio, lactate dehydrogenase, blood routine, schistocytes will be detected at regular times.
2. According to the diagnostic criteria of TA-TMA, TA-TMA patients and 1:1 matched non-TA-TMA patients will be screened, and the training set (30 cases each) and validation set (10 cases each) will be established respectively. Plasma warning biomarkers with high sensitivity, stability, and accuracy will be screened and identified from the large amount of data by proteomics and metabolomics technologies.
3. intending to utilize the opportunity of this clinical study to collect clinical data and biological samples from allo-HSCT patients, establish a clinical database and biological samples bank for TA-TMA disease, and provide sample support for subsequent translational research.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosis of a hematologic disease (e.g., leukemia, myelodysplastic syndromes,lymphoma) confirmed by histology or other appropriate diagnostic methods.
* 2. undergoing allo-HSCT
* 3. Age 14 years or older
* 4.Informed consent must be signed before the start of the study. For participants aged 18 and above, the informed consent should be signed by the patient or their immediate family member. Considering the patient's condition, if it is not favorable for the patient to sign, the informed consent may be signed by a legal guardian or immediate family member of the patient.

Exclusion Criteria:

* 1. Missing or lost follow-up of key clinical data
* 2. failure to collect plasma samples at specific time points after transplantation
* 3. Plasma sample collection time later than the onset date of TMA
* 4. TMA occurrence time later than 180 days after transplantation

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include patients aged 14 years and older who have undergone allogeneic hematopoietic stem cell transplantation for hematologic disorders. Complement, blood smear, renal function, and complete blood count tests at specified time points will be conducted to assess the patients' health status. The investigators anticipate enrolling a minimum of 300 patients and will calculate the incidence rate of TA-TMA according to international diagnostic standards.Based on subsequent occurrences of TATMA in patients, the study population will be categorized into two groups: the TATMA occurrence group and the non-TATMA occurrence group.The objective of this study is to gain insights into the potential role of complement testing in TA-TMA
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
plasma biomarkers to predict TA-TMA | from transplantation to the onset of TATMA
  By matching the TMA group with the control group, we aim to identify plasma biomarkers that can predict the early onset of TMA.
the survival of patients with TATMA | 1-year after transplantation
  the 1-year OS of patients with TATMA

SECONDARY OUTCOMES:
non-relapse mortality | one or two years after transplantation
  the non-relapse mortality for patients

CONTACTS AND LOCATIONS:
Overall Officials: Erlie Jiang, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, China